CLINICAL TRIAL: NCT02149771
Title: Transarterial Chemoembolisation (TACE) Combined With Endovascular Implantation of Bare Stent and Iodine-125 Seed Strand for the Treatment of Hepatocellular Carcinoma With Portal Vein Tumour Thrombosis Versus TACE Alone
Brief Title: Combination Treatment for Advanced Liver Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Zhiping Yan, Prof., Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR 2013
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma; Hepatic Portal Vein Tumor Invasion
Keywords: hepatocellular carcinoma; portal vein tumor thrombosis; stents; chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TACE&Stents (Experimental): chemoembolization combined with endovascular stents and iodine-125 seed strand implantation
  Interventions: Procedure: chemoembolization; Device: endovascular stents implantation; Procedure: iodine-125 seed strand implantation
- TACE (Active Comparator): Transartery chemoembolisation（TACE） by administering Doxorubicin and Oxaliplatin mixed with 5-20 mL iodised oil.Gelatine sponge was used to embolise the feeding artery of the tumour.Repeat if patients with viable lesions demonstrated by CT or MRI.
  Interventions: Procedure: chemoembolization

INTERVENTIONS:
Procedure: chemoembolization — Conventional chemoembolisation by administering Doxorubicin and Oxaliplatin mix with 5-20 mL iodised oil.Gelatine sponge was used to embolise the feeding artery of the tumour.Repeat if patients with viable lesions demonstrated by CT or MRI.
Device: endovascular stents implantation — Bare stents implant within portal vein.
  Arms: TACE&Stents
Procedure: iodine-125 seed strand implantation — Iodine-125 seed strand implant within portal vein.
  Arms: TACE&Stents

SUMMARY:
The purpose of this study is to determine whether TACE combined endovascular stent implantation confers a survival benefit over TACE alone.

ELIGIBILITY:
Inclusion Criteria:

* (1) Hepatocellular carcinoma(HCC) diagnosis confirmed by needle biopsy or by two coincidental imaging techniques associated with increased α-fetoprotein according to the American Association for the Study of Liver Diseases (AASLD) guidelines and contrast-enhancing tumour thrombus within the main portal vein and one of the first-order branch on CT or MRI;
* (2) Child-Pugh classification grade A or B；
* （3）Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less.

Exclusion Criteria:

* advanced liver disease (bilirubin levels >3 mg/dL, ASTor ALT >5 × upper limit of normal)；
* Tumor invade the Inferior Vena Cava, extrahepatic spread;
* contraindications for doxorubicin or oxaliplatin chemotherapy;
* any contraindication to an arterial procedure such as impaired clotting tests (platelet count below 50 × 109/L or prothrombin activity below 50 %);
* renal failure,cardiac ejection fraction <50 %) or end-stage disease；
* patients who were not capable of cooperation during the procedure.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Median survival time | 2 years

SECONDARY OUTCOMES:
Time to Disease Progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhinping Yan, MD, Principal Investigator — Department of Interventional Radiology, Zhongshan Hospital, Fudan University; Jianjun Luo, MD, Study Director — Department of Interventional Radiology, Zhongshan Hospital, Fudan University
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China